CLINICAL TRIAL: NCT05484427
Title: Kids Diabetes Telemedicine Study (KITES)
Acronym: KITES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Lenka Petruzelkova, Principle investigator - Lenka Petruzelkova, MD, PhD., University Hospital, Motol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-CIP-24-02-2021
Record Dates: First submitted 2021-04-27; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes children; Telemedicine; Virtual clinic
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Randomised prospective single-center trial
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine arm (Experimental): Participants in this arm will be follow up by telemedicine control (via emails) instead of regular controls. They will upload the data from their devices (pump, CGM) to cloud system on their own. All instructions what to change they will recive by email only.
  Interventions: Other: Telemedicine
- Outpatient clinic meetings arm (No Intervention): Participants in this arm will normally come for the regular meetings with their diabetologist to the outpatient clinic.

INTERVENTIONS:
Other: Telemedicine — Replacement of the regullar meeting with diabetologist by remote communication only
  Arms: Telemedicine arm

SUMMARY:
Randomised prospective single-center clinical trial evaluating the outcomes of children with type 1 diabetes followed up by remote telemedicine check-ups without their personal present at the outpatient clinic.

DETAILED DESCRIPTION:
At the first study visit (visit Month 0), after obtaining the written informed consent from the parents, 50 children with type 1 diabetes will be randomised to two groups of equal size.

The first group will have regular visits with their diabetologist to our outpatient clinic every 3 months (visits Month 3 and Month 6), the second group will have a remote control by email only instead of regular visits (visits Month 3 and Month 6). The CGM data and inzulin dose will be evaluated through cloud systems (Diasend, Carelink) at every control by diabetologist. The patients would be instructed about the reccomendation during the "live" control or by email according the group. The final meeting (visit Month 9) will take place at our outpatient clinic for both of the study groups. The CGM data, HbA1c, and the questionaire evaluating the quality of the controls will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes
* Age 1-18 years
* Type 1 diabetes duration at least 12 months
* Using continuous glucose monitoring for at least previous 6 months
* Willingness to use continuous glucose monitoring for the whole study
* Signed informed consent by the legal representatives

Exclusion Criteria:

* Change of the type 1 treatment modalitry (from insulin pens to insulin pump or vice versa, start the treatment with hybrid closed loop, start of the treatment with the drug affecting the glucose metabolism) in 3 months prior to the study or planning to change the treatment modality during the study
* Concomitant psychiatric diagnosis diagnosed by the psychiatrist
* Hospitalisation for severe hypoglycaemia and/or diabetic ketoacidosis in 1 year prior to the study initiation
* Glycated hemoglobin concentration >90 mmol/mol in 1 year prior to the study or substantially bad co-operation of the patient/parent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
metabolic control (HbA1c concentrations) at Month 9 | Month 9 visit
  The noninferiority of HbA1C concentration between the groups (the difference of HbA1c between the groups will be less than 5 mmol/mol,

SECONDARY OUTCOMES:
Control of glycemia levels by CGM data evaluation. | Month 3, Month 6, and Month 9
  To compare the CGM data (time in range, hypoglyceamia, hyperglycaemia, SD, ...) between the groups.
Duration of the dia visit | Month 3and Month 6
  To compare the time duration of dia visit between the groups. The time duration of each visits will be measured by doctor and patient separately.
  Doctor´s and patient´s time duration of the visits will be compared
Patient´s satisfaction of regular and telemedicine (email) visits. | Month 9
  Patient´s satisfaction of regular and telemedicine (email) visits wil be compared by special questionnare.

CONTACTS AND LOCATIONS:
Overall Officials: Lenka Petruzelkova, MD, PhD., Principal Investigator — Motol University Hospital
Locations (1):
- Department of Paediatrics, Motol University Hospital 2nd Medical Faculty in Prague, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the anonymised participants' data on individual request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after study termination, for 2 years time

REFERENCES:
- [Derived] Plachy L, Neuman V, Velichova K, Slavenko MG, Santova A, Anne Amaratunga S, Obermannova B, Kolouskova S, Pruhova S, Sumnik Z, Petruzelkova L. Telemedicine maintains good glucose control in children with type 1 diabetes but is not time saving for healthcare professionals: KITES randomized study. Diabetes Res Clin Pract. 2024 Mar;209:111602. doi: 10.1016/j.diabres.2024.111602. Epub 2024 Mar 2. PMID 38437986